CLINICAL TRIAL: NCT03762317
Title: Clonidine as Adjunct to Morphine in the Management of Term and Near Term Infants With Neonatal Abstinence Syndrome
Brief Title: Clonidine as Adjunct to Morphine for Neonatal Abstinence Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was initially suspended due to IND application and later terminated due to the difficulty of obtaining consent during COVID period
Sponsor: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Principal Investigator, kunal gupta, Assistant Professor, Hennepin County Medical Center, Minneapolis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAS
Record Dates: First submitted 2017-11-08; First posted 2018-12-03 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- clonidine (Active Comparator): Clonidine is started at 6mcg/kg/day and increased to 12 mcg/kg/d for the duration of the study period
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator): Placebo solution will be given for the duration of the study period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — clonidine will be given at 12 mcg/kg/d to the experimental arm in addition to oral morphine
  Arms: clonidine
Drug: Placebo — Placebo with volume similar to clonidine at 12 mcg/kg/d will be given to this arm in addition to oral morphine
  Arms: Placebo

SUMMARY:
This is a prospective randomized double blinded study comparing the effect on duration of pharmacologic treatment and duration of hospital stay when using clonidine at 12 µg/kilogram/day as an adjunct to oral morphine as compared to morphine monotherapy in the management of term and near term infants with neonatal abstinence syndrome (NAS)

DETAILED DESCRIPTION:
Neonatal abstinence syndrome (NAS) is an emerging epidemic and has lead to a tremendous increase in cost of medical care. Opioids are the mainstay of treatment for NAS although there are concerns about possible short-term and long-term effects including but not limited to adverse neurodevelopmental outcomes. Other drugs such as clonidine, phenobarbitone, methadone and buprenorphine have been evaluated to limit the postnatal exposure to opioids in these infants. Clonidine is an alpha 2 receptor and can lessen withdrawal manifestations. The addition of clonidine at 6 µg/kilogram/day to morphine in the management of NAS has been shown to reduce the duration of pharmacotherapy by about 27% in a previous study.

A recent pilot study reported reduction of treatment duration for NAS with clonidine (12 µg/kilogram/day) monotherapy as compared to morphine monotherapy. The study reported no adverse effects in study subjects at the doses used in the study. The investigators hypothesize that there will be a minimum of 30% reduction in the treatment duration with 12 µg/kilogram/day clonidine used as adjuncts to standard morphine treatment as compared to morphine monotherapy in the management of term and near term infants with NAS

ELIGIBILITY:
Inclusion Criteria:

* Requiring neonatal intensive care unit (NICU) admission for management of neonatal abstinence syndrome
* Gestational age greater than or equal to 36 weeks
* Less than or equal to 48 hours of treatment with morphine for NAS

Exclusion Criteria:

* Presence of seizures
* Congenital malformations, genetic syndromes or the presence of TORCH infections
* Major medical problems
* Heart rate and/or blood pressure instability

Ages: 36 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: kunal gupta, Principal Investigator — Hennepin County Medical Center, Minneapolis; vinay sharma, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized blinded study where the HCMC research pharmacist assigned the randomization group and provided the study medication and placebo
Period: Overall Study
Arm/Group | Clonidine | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: weeks] | 39 [37.3 to 42] | 37.4 [36 to 39.1] | 38.3 [36 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Duration of Pharmacotherapy for NAS
Description: The length of time in days from the initiation of pharmacotherapy on day 1 until the medication has been stopped
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
days | 30.2 (18.6) | 25.6 (14.7)

2. Secondary Outcome: Duration of Hospital Stay
Description: Number of days spent in the hospital
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
days | 32.4 (17.3) | 31.6 (13.4)

3. Secondary Outcome: Maximum Dose of Morphine Used
Description: The maximum dose of morphine in mg/kg used for symptom control
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
mg/kg | 0.11 (0.05) | 0.10 (0.03)

4. Secondary Outcome: Average Daily Dose of Oral Morphine Over Hospital Stay
Description: The average daily dose of morphine used throughout study period in mg/kg/day
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
mg/kg/day | 0.4 (0.2) | 0.4 (0.2)

5. Secondary Outcome: Total Number of Episodes of Heart Rate Variability (Heart Beats/Min)
Description: Number of episodes of bradycardia (Heart rate < 60/min for a minimum of 20 seconds and not associated with apnea or signs of reflux such as emesis, regurgitation of milk into the mouth or nose, arching while feeding, number of episodes of tachycardia (Heart rate > 200/min) and not related to pain and/or agitation
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Number; unit: events
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
events | 0 | 0

6. Secondary Outcome: Total Number of Episodes of Blood Pressure (mm of Hg) Variability
Description: Number of episodes of hypotension (blood pressure < 5th percentile for age) and hypertension (blood pressure > 95th percentile for age)
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Measure: Number; unit: episodes
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 5 | 5
episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: From beginning of morphine therapy during NICU admission until discharge from the hospital, up to 100 days
Arm/Group | Clonidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03762317/Prot_SAP_001.pdf